CLINICAL TRIAL: NCT04409327
Title: Randomized Double Blind Placebo-Controlled Study to Determine if Prophylaxis With RTB101 Compared to Placebo Reduces Severity of Lab Confirmed COVID19 in Adults ≥65 Years in a Nursing Home in Which ≥1 Person(s) Have Lab Confirmed COVID19
Brief Title: Phase 2 Study to Determine if RTB101 Reduces the Severity of COVID-19 in Older Adults Residing in Nursing Homes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient accrual rate
Sponsor: Restorbio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RTB101-210
Record Dates: First submitted 2020-05-28; First posted 2020-06-01 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: COVID19
Keywords: Mechanistic Target of Rapamycin (mTOR); Virus
MeSH Terms: conditions — COVID-19; Hereditary Sensory and Autonomic Neuropathies; Virus Diseases | interventions — dactolisib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 10 mg daily RTB101 (Experimental): TORC1 inhibitor
  Interventions: Drug: RTB101
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RTB101 — Oral RTB101 10 mg hard gelatin capsule once daily for 4 weeks
  Other Names: Dactolisib; BEZ235
  Arms: 10 mg daily RTB101
Drug: Placebo — Oral matching placebo once daily for 4 weeks
  Other Names: Placebo capsule
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if prophylaxis with RTB101 decreases the severity of laboratory-confirmed COVID-19 among adults ≥ 65 years who reside in a nursing homes in which one or more residents or staff have laboratory-confirmed COVID-19

DETAILED DESCRIPTION:
RTB101-210 is Placebo-Controlled Study to Determine if Prophylaxis with RTB101 as Compared to Placebo Reduces the Severity of Laboratory-Confirmed COVID-19 in Adults Age ≥65 Years who Reside in a Nursing Home in which One or More Residents or Staff have Laboratory-Confirmed COVID-19. This trial is being conducted in follow up to a Phase 3 trial, in which trends toward a reduction in the severity of laboratory-confirmed RTIs including coronavirus RTIs were again seen. Therefore, RTB101 is a potential pan antiviral immunotherapy that may prevent or ameliorate viral RTIs, including COVID-19, in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent must be obtained from the subject or health care proxy before any assessment is performed.
* Adults (male and female) aged 65 years and over.
* Residing in a nursing home in which one or more residents or staff has developed laboratory-confirmed symptomatic COVID-19 infection at the time of randomization

Exclusion Criteria:

Subjects will not be eligible if they meet any of the following criteria:

* Any subject who is a current smoker or has a ≥ 10 pack year smoking history.
* Subjects with a medical history of chronic obstructive pulmonary disease (COPD).
* Subjects who are in hospice or receiving comfort care only.
* Subjects who have symptomatic laboratory-confirmed COVID-19 at the time of screening or randomization.
* Subjects with current evidence of an unstable medical disorder including an unstable respiratory disorder, gastrointestinal disorder (including Child-Pugh class B and C hepatic impairment), renal disorder (including subjects with an estimated glomerular filtration rate (eGFR) ≤30 mL/min/1.73m2), or hematologic disorder (including active leukemia).
* Subjects receiving immunosuppressive therapy including chronic use of prednisone >10 mg daily (however, inhaled corticosteroids and acute use of higher doses of prednisone to treat conditions such as exacerbation of asthma or other acute conditions are allowed).
* Subjects with an immunodeficiency disease, including a positive human immunodeficiency virus (HIV) test result.
* Sexually active males with a partner of child-bearing potential

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-07-11 (Actual); Primary Completion 2020-12-27 (Actual); Study Completion 2021-01-24 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects who develop laboratory-confirmed COVID-19: - with protocol-defined progressive symptoms OR - are hospitalized OR - die | Through Week 4

SECONDARY OUTCOMES:
The percentage of subjects who develop symptomatic laboratory-confirmed COVID-19 infection | Through Week 4
Mortality rate in subjects who develop laboratory-confirmed COVID19 | Through Week 8
Percent of subjects who are hospitalized due to having one or more predefined COVID-19 symptoms and laboratory-confirmed SARS-CoV-2 | Through Week 4
Percent of subjects who require mechanical ventilation, noninvasive ventilation, high flow nasal canula oxygen delivery or ICU admission during the hospitalization for COVID19 | Through Week 8
Safety and tolerability will be assessed by report of AE/SAEs | Through Week 5 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Restorbio Inc.
Locations (1):
- Nursing Home, Middletown, Rhode Island, United States